CLINICAL TRIAL: NCT01610336
Title: A Phase IB/II, Open Label, Multicenter Study of INC280 Administered Orally in Combination With Gefitinib in Adult Patients With EGFR Mutated, c-MET-amplified Non-small Cell Lung Cancer Who Have Progressed After EGFR Inhibitor Treatment
Brief Title: A Safety and Efficacy Study of INC280 and Gefitinib in Patients With EGFR Mutated, c-MET-amplified NSCLC Who Have Progressed After EGFRi Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINC280X2202; 2011-002569-39 (EudraCT Number)
Record Dates: First submitted 2012-04-03; First posted 2012-06-04 (Estimated); Results first posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: EGFR; c-MET; Lung cancer; Gefitinib; Erlotinib; Non-small cell lung cancer (NSCLC); lung adenocarcinoma; large-cell lung carcinoma
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Adenocarcinoma of Lung | interventions — capmatinib; Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (11):
- INC280 100 mg Cap QD Phase Ib (Experimental): cap=capsule; QD=once daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 200 mg Cap QD Phase Ib (Experimental): cap=capsule; QD=once daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 400 mg Cap QD Phase Ib (Experimental): cap=capsule; QD=once daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 800 mg Cap QD Phase Ib (Experimental): cap=capsule; QD=once daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 200 mg Cap BID Phase Ib (Experimental): cap=capsule; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 400 mg Cap BID Phase Ib (Experimental): cap=capsule; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 600 mg Cap BID Phase Ib (Experimental): cap=capsule; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 200 mg Tab BID Phase Ib (Experimental): tab=tablet; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 400 mg Tab BID Phase Ib (Experimental): tab=tablet; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 400 mg Cap BID Phase II (Experimental): cap=capsule; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib
- INC280 400 mg Tab BID Phase II (Experimental): tab=tablet; BID=twice daily
  Interventions: Drug: INC280; Drug: Gefitinib

INTERVENTIONS:
Drug: INC280 — During Phase Ib, INC280 was taken at escalating doses. During Phase II part, INC280 was taken at recommended Phase II dose.
  Other Names: Capmatinib
Drug: Gefitinib — Gefitinib 250 mg taken once daily

SUMMARY:
This study assessed the safety and efficacy of escalating doses INC280 when added to gefitinib in patients with lung cancer that were known to have dysregulation of the c-MET pathway and who had failed after benefiting on a prior treatment with either gefitinib or erlotinib.

DETAILED DESCRIPTION:
The Phase Ib dose escalation part was aimed at the determination of the MTD/RP2D of capmatinib in combination with 250 mg gefitinib in patients with NSCLC patients with epidermal growth factor receptor (EGFR) mutation and cMET dysregulation and showing disease progression following EGFR tyrosine-kinase inhibitor (EGFR TKI) therapy. Dose escalation started with a dose of 100 mg/day to a maximum of 1200 mg/day, as capsule or tablet formulation. Successive cohorts of patients were to receive increasing doses of capmatinib in combination with a 250 mg once daily (qd) dose of gefitinib until the MTD/RP2D of capmatinib had been determined. The Phase II dose expansion part consisted of 400 mg capmatinib twice daily (bid), as either capsules or tablets, in combination with 250 mg gefitinib.

ELIGIBILITY:
Inclusion Criteria:

* Documented EGFR mutation
* Documented c-MET dysregulation
* Prior clinical benefit on EGFR inhibitors and then subsequent progression

  -≥ 18 year old
* Life expectancy of ≥ 3 months
* ECOG performance status ≤ 2

Exclusion Criteria:

* Unable to swallow tables once or twice daily
* Previous treatment with c-MET inhibitor
* Any unresolved toxicity from previous anticancer therapy greater than grade 1
* History of cystic fibrosis
* History of acute or chronic pancreatitis
* Unable to undergo MRI or CT scans
* Known history of HIV
* Undergone a bone marrow or solid organ transplant
* Clinically significant wound or lung tumor lesions with increased likelihood of bleeding
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 161 (Actual)
Dates: Start 2012-04-05 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (29):
- Australia (3):
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, East Bentleigh, Victoria
  - Novartis Investigative Site, Auckland
- Novartis Investigative Site, Leuven, Belgium
- China (4):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Shanghai, Shanghai Municipality
  - Novartis Investigative Site, Beijing
  - Novartis Investigative Site, Guangzhou
- France (2):
  - Novartis Investigative Site, Strasbourg
  - Novartis Investigative Site, Toulouse
- Germany (2):
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Freiburg im Breisgau
- Novartis Investigative Site, Ramat Gan, Israel
- Italy (2):
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Modena, MO
- Novartis Investigative Site, Koto Ku, Tokyo, Japan
- Netherlands (3):
  - Novartis Investigative Site, Maastricht, AZ
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Singapore, Singapore
- South Korea (4):
  - Novartis Investigative Site, Gyeonggi-do, Korea
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho Gu
  - Novartis Investigative Site, Seoul
- Spain (2):
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, Madrid
- Taiwan (2):
  - Novartis Investigative Site, Tainan
  - Novartis Investigative Site, Taipei
- Novartis Investigative Site, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Wu YL, Zhang L, Kim DW, Liu X, Lee DH, Yang JC, Ahn MJ, Vansteenkiste JF, Su WC, Felip E, Chia V, Glaser S, Pultar P, Zhao S, Peng B, Akimov M, Tan DSW. Phase Ib/II Study of Capmatinib (INC280) Plus Gefitinib After Failure of Epidermal Growth Factor Receptor (EGFR) Inhibitor Therapy in Patients With EGFR-Mutated, MET Factor-Dysregulated Non-Small-Cell Lung Cancer. J Clin Oncol. 2018 Nov 1;36(31):3101-3109. doi: 10.1200/JCO.2018.77.7326. Epub 2018 Aug 29. PMID 30156984

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Started | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Not completed — Progressive Disease | 4 | 6 | 6 | 5 | 3 | 10 | 1 | 6 | 6 | 40 | 36
Not completed — Adverse Event | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 2 | 8 | 6
Not completed — Subject/Guardian decision | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 2 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 1 | 2
Not completed — Non-Compliance with study treatment | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Deviation | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Transfer to another trial | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II | Total
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.8 (11.05) | 60.4 (15.27) | 59.5 (6.89) | 51.3 (8.88) | 64.5 (8.89) | 55.9 (10.81) | 61.0 (8.46) | 60.9 (12.86) | 58.4 (5.01) | 58.6 (10.50) | 62.8 (9.32) | 59.7 (10.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 4 | 5 | 4 | 4 | 2 | 5 | 5 | 33 | 19 | 88
  Male | 3 | 2 | 2 | 2 | 0 | 8 | 3 | 2 | 3 | 20 | 28 | 73
Race/Ethnicity, Customized [Number; unit: Participants]
  Russian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Mixed Ethnicity | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Not reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 3
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 5 | 7
  Southeast Asian | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 8 | 12
  Other | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 0 | 11 | 17
  East Asian | 4 | 6 | 6 | 7 | 3 | 9 | 4 | 3 | 7 | 53 | 16 | 118

OUTCOME MEASURES:

1. Primary Outcome: Phase Ib: Frequency of Dose Limiting Toxicities (DLTs)
Description: A dose-limiting toxicity (DLT) was defined as an adverse event or abnormal laboratory value assessed as unrelated to disease progression, inter-current illness, or concomitant medications that met certain criteria as defined in the protocol.
Time Frame: Up to 215 weeks
Population: Safety Set: All patients in phase Ib who received at least one full or partial dose of INC280 or gefitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 3 | 7 | 6 | 5 | 4 | 10 | 1 | 7 | 7
Participants
  Cough | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Dizziness | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Dyspnoea | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Phase II : Overall Response Rate (ORR)
Description: Overall response rate is defined as the proportion of patients with best overall response (BOR) of complete response (CR) or partial response (PR), as per RECIST 1.1 (Overall Response (OR) = CR + PR).
  Complete Response (CR): Disappearance of all non-nodal target lesions. In addition, any pathological lymph nodes assigned as target lesions must have a reduction in short axis to < 10 mm Partial Response (PR): At least a 30% decrease in the sum of diameter of all target lesions, taking as reference the baseline sum of diameters.
Time Frame: Until disease progression, up to 60.8 weeks
Population: Full analysis set: all patients in phase II who receive at least one full or partial dose of INC280 or gefitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 53 | 47
Participants | 12 | 17

3. Secondary Outcome: Phase Ib and II: Number of Participants With Adverse Events (AEs)
Description: Adverse events were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 421 weeks
Population: Safety Set: All patients in phase Ib and II who received at least one full or partial dose of INC280 or gefitinib and and had at least one valid postbaseline safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Participants
  AEs | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 51 | 47
  Grade 3/4 AEs | 3 | 4 | 2 | 4 | 2 | 6 | 4 | 6 | 4 | 24 | 35

4. Secondary Outcome: Phase Ib and II: Number of Participants With Serious Adverse Events (SAEs)
Description: Serious adverse events were assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0
Time Frame: Up to 421 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Participants | 1 | 2 | 2 | 3 | 0 | 4 | 3 | 5 | 3 | 12 | 19

5. Secondary Outcome: Phase Ib and II: Number of Patients With Dose Reductions of INC280 by Dose Level
Description: Number of patients with dose reductions of INC280 by dose level as a measure of tolerability.
Time Frame: Up to 417 weeks
Population: Safety Set: All patients in phase Ib and II who received at least one full or partial dose of INC280 or gefitinib.
Measure: Count of Participants; unit: Participants
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Participants
  Without dose reductions | 5 | 6 | 5 | 6 | 1 | 8 | 1 | 5 | 5 | 30 | 23
  Only 1 dose reduction | 0 | 1 | 0 | 1 | 2 | 2 | 2 | 0 | 1 | 13 | 17
  2 dose reductions | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 1 | 1 | 6 | 5
  3 dose reductions | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 1
  >3 dose reductions | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 3 | 1

6. Secondary Outcome: Phase Ib and II: Number of Patients With Dose Interruptions of Gefitinib by Dose Level
Description: Number of patients with dose interruptions of gefitinib by dose level as a measure of tolerability
Time Frame: Up to 417 weeks
Population: Safety set: All patients in phase Ib and II who received at least one full or partial dose of INC280 or gefitinib.
Measure: Count of Participants; unit: Participants
Groups:
- mg Cap BID Phase II: cap=capsule; BID=twice daily
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 5 | 7 | 6 | 7 | 4 | 12 | 5 | 7 | 8 | 53 | 47
Participants
  Without dose interruptions | 5 | 5 | 6 | 4 | 4 | 6 | 4 | 4 | 4 | 42 | 25
  With only one dose interruption | 0 | 2 | 0 | 2 | 0 | 3 | 0 | 0 | 2 | 9 | 16
  2 dose interruptions | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 4
  3 dose interruptions | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 2
  >3 dose interruptions | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0

7. Secondary Outcome: Phase II: Overall Survival (OS)
Description: Overall survival is defined as the time from the start of treatment date to the date of death, due to any cause
Time Frame: From date of treatment until death due to any cause, up to 70.2 months
Population: Full analysis set: all patients in phase II who receive at least one full or partial dose of INC280 or gefitinib.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 53 | 47
Months | 12.3 [8.1 to 15.4] | 15.2 [11.7 to 20.1]

8. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: Progression-free survivalis the time from date of randomization/start of treatment to the date of event defined as the first documented progression or death due to any cause.
Time Frame: Up to 60.8 months
Population: Full analysis set: all patients in phase II who receive at least one full or partial dose of INC280 or gefitinib
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 53 | 47
Months | 5.1 [3.6 to 5.6] | 5.5 [3.8 to 7.3]

9. Secondary Outcome: Phase II: Duration of Response (DoR)
Description: Duration of overall response (DOR) is defined as the time between the date of first documented response (CR or PR) and the date of first documented disease progression or death due to underlying cancer.
Time Frame: Up to 23.2 months
Population: Full analysis set subjects in phase II with confirmed complete response (CR) or partial response (PR)
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 12 | 17
Months | 5.6 [3.7 to 6.2] | 5.6 [3.7 to 7.4]

10. Secondary Outcome: Phase I: PK Parameters AUCtau of INC280 and Gefitinib
Description: PK parameters were estimated from each individual plasma concentration-time profile using non-compartmental analysis.
  Area under the plasma concentration-time curve (AUC) from time zero to the end of dosing interval at steady state (tau), where tau=24 hours for once daily dosing and tau=12 hours for twice daily dosing
Time Frame: Cycle 1 day 15 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose) (Cycle=28 days)
Population: Pharmacokinetic analysis set: all patients having at least one evaluable PK profile of INC280 and/or gefitinib. Patients were included on the estimation of this PK parameter if a sufficient number of blood samples was available.
Measure: Mean (Standard Deviation); unit: hr∙ng/mL
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 4 | 7 | 5 | 3 | 4 | 10 | 2 | 7 | 7
hr∙ng/mL
  INC280 | 4510 (1960) | 9140 (5550) | 29200 (12700) | 30300 (19800) | 9660 (5780) | 21400 (8420) | 37300 (18800) | 13900 (4470) | 28700 (5460)
  Gefitinib: number analyzed (Participants) | 3 | 6 | 3 | 1 | 2 | 6 | 0 | 5 | 4
  Gefitinib | 7690 (1400) | 8070 (2080) | 7140 (1830) | 12800 | 8440 (2360) | 8500 (5330) |  | 7160 (2040) | 7820 (1130)

11. Secondary Outcome: Phase I: PK Parameters Cmax of INC280 and Gefitinib
Description: PK parameters were estimated from each individual plasma concentration-time profile using non-compartmental analysis.
  Cmax is the maximum observed plasma concentration of INC280 and gefitinib
Time Frame: Cycle 1 day 15 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose) (Cycle=28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 4 | 7 | 6 | 4 | 4 | 10 | 2 | 7 | 7
ng/mL
  INC280 | 826 (521) | 1490 (1430) | 4620 (3060) | 6570 (4360) | 1950 (985) | 4220 (2100) | 4840 (1990) | 2550 (676) | 6760 (1740)
  Gefitinib | 417 (42.9) | 378 (85.2) | 405 (144) | 357 (225) | 480 (191) | 464 (209) | 255 (158) | 479 (167) | 355 (74.1)

12. Secondary Outcome: Phase I: PK Parameters Tmax of INC280 and Gefitinib
Description: PK parameters were estimated from each individual plasma concentration-time profile using non-compartmental analysis.
  Tmax is the time to reach maximum plasma concentration of INC280 and gefitinib
Time Frame: Cycle 1 day 15 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose) (Cycle=28 days)
Population: as for outcome 10
Measure: Median (Full Range); unit: Hours
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 4 | 7 | 6 | 4 | 4 | 10 | 2 | 7 | 7
Hours
  INC280 | 1.96 [1.50 to 3.92] | 2.00 [1.00 to 24.0] | 2.00 [1.98 to 6.00] | 2.05 [1.92 to 5.97] | 1.50 [1.00 to 3.98] | 2.00 [0.50 to 4.00] | 5.00 [4.00 to 6.00] | 2.00 [1.00 to 4.00] | 1.08 [1.00 to 4.00]
  Gefitinib | 3.92 [0 to 8.00] | 6.00 [3.97 to 24.0] | 6.02 [2.00 to 8.0] | 5.94 [2.10 to 7.28] | 5.00 [4.00 to 8.00] | 6.00 [3.97 to 8.00] | 11.3 [0 to 22.5] | 6.00 [2.00 to 7.50] | 6.00 [3.90 to 7.95]

13. Secondary Outcome: Phase I: PK Parameters Apparent Systemic Plasma Clearance Rate of INC280 and Gefitinib
Description: PK parameters were estimated from each individual plasma concentration-time profile using non-compartmental analysis.
  Apparent systemic plasma clearance rate of INC280 and gefitinib
Time Frame: Cycle 1 day 15 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose) (Cycle=28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 4 | 7 | 5 | 3 | 4 | 10 | 2 | 7 | 7
L/hr
  INC 280 | 26.9 (15.0) | 29.4 (15.7) | 16.3 (7.61) | 47.7 (49.1) | 27.0 (14.7) | 24.2 (18.3) | 18.4 (9.31) | 15.4 (3.89) | 14.4 (3.10)
  Gefitinib: number analyzed (Participants) | 3 | 6 | 3 | 1 | 2 | 6 | 0 | 5 | 4
  Gefitinib | 33.3 (6.78) | 32.9 (9.65) | 36.5 (8.41) | 19.5 | 30.8 (8.61) | 41.0 (24.1) |  | 36.9 (8.81) | 32.5 (4.99)

14. Secondary Outcome: Phase I: PK Parameters Half-life of INC280 and Gefitinib
Description: PK parameters were estimated from each individual plasma concentration-time profile using non-compartmental analysis.
  The elimination half-life of INC280 and gefitinib associated with the terminal slope (Lamda_z) of a semi-logarithmic plasma concentration-time curve
Time Frame: Cycle 1 day 15 (pre-dose, 0.5, 1, 2, 4, 6, 8 and 24 hours post dose)(Cycle=28 days)
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib
Number analyzed (Participants) | 4 | 6 | 5 | 3 | 3 | 9 | 0 | 7 | 6
hours
  INC280 | 3.86 (0.564) | 5.10 (2.01) | 3.16 (0.361) | 3.67 (0.796) | 3.19 (0.942) | 3.01 (1.38) |  | 3.75 (1.94) | 3.17 (0.783)
  Gefitinib: number analyzed (Participants) | 1 | 3 | 2 | 1 | 2 | 3 | 0 | 3 | 1
  Gefitinib | 18.8 | 26.9 (4.63) | 36.3 (8.20) | 37.8 | 16.3 (2.16) | 18.7 (7.75) |  | 17.8 (5.08) | 23.9

15. Other Pre Specified Outcome: Phase I: Percentage of Change From Baseline in C-MET H Score at Cycle 1 Day 15
Description: Inhibition of c-MET signaling by pre- and post- treatment immunohistochemistry of p-c-MET
Time Frame: Baseline, Day 15 of cycle 1 (Cycle=28days)
Population: Full analysis set patients in phase Ib with p cMET H score measured. Few tumor samples were available since tumor biopsy was optional for this study.
Measure: Median (Full Range); unit: Percentage
Arm/Group | INC280 100 mg Cap QD Phase Ib | INC280 200 mg Cap QD Phase Ib | INC280 400 mg Cap QD Phase Ib | INC280 800 mg Cap QD Phase Ib | INC280 200 mg Cap BID Phase Ib | INC280 400 mg Cap BID Phase Ib | INC280 600 mg Cap BID Phase Ib | INC280 200 mg Tab BID Phase Ib | INC280 400 mg Tab BID Phase Ib | INC280 400 mg Cap BID Phase II | INC280 400 mg Tab BID Phase II
Number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Percentage | -100 [-100 to -100] |  |  |  |  | -100 [-100 to -100] |  |  |  | -31 [-31 to -31] |

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment plus 30 days post treatment, up to maximum duration of 8 years.
Description: Any sign or symptom that occurs during the study treatment plus the 30 days post treatment.
Groups:
- 100 mg Cap QD (Ph Ib): 100 mg Cap QD (Ph Ib)
- 200 mg Cap QD (Ph Ib): 200 mg Cap QD (Ph Ib)
- 400 mg Cap QD (Ph Ib): 400 mg Cap QD (Ph Ib)
- 800 mg Cap QD (Ph Ib): 800 mg Cap QD (Ph Ib)
- 200 mg Cap BID (Ph Ib): 200 mg Cap BID (Ph Ib)
- 400 mg Cap BID (Ph Ib): 400 mg Cap BID (Ph Ib)
- 600 mg Cap BID (Ph Ib): 600 mg Cap BID (Ph Ib)
- 200 mg Tab BID (Ph Ib): 200 mg Tab BID (Ph Ib)
- 400 mg Tab BID (Ph Ib): 400 mg Tab BID (Ph Ib)
- 400 mg Cap BID (Ph II): 400 mg Cap BID (Ph II)
- 400 mg Tab BID (Ph II): 400 mg Tab BID (Ph II)
Arm/Group | 100 mg Cap QD (Ph Ib) | 200 mg Cap QD (Ph Ib) | 400 mg Cap QD (Ph Ib) | 800 mg Cap QD (Ph Ib) | 200 mg Cap BID (Ph Ib) | 400 mg Cap BID (Ph Ib) | 600 mg Cap BID (Ph Ib) | 200 mg Tab BID (Ph Ib) | 400 mg Tab BID (Ph Ib) | 400 mg Cap BID (Ph II) | 400 mg Tab BID (Ph II)
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/7 | 0/6 | 1/7 | 0/4 | 1/12 | 3/5 | 0/7 | 1/8 | 6/53 | 2/47
Serious Adverse Events (participants affected / at risk) | 1/5 | 2/7 | 2/6 | 3/7 | 0/4 | 4/12 | 3/5 | 5/7 | 3/8 | 12/53 | 19/47
Other Adverse Events (participants affected / at risk) | 5/5 | 7/7 | 6/6 | 7/7 | 4/4 | 12/12 | 4/5 | 6/7 | 7/8 | 49/53 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Cap QD (Ph Ib) (N=5) | 200 mg Cap QD (Ph Ib) (N=7) | 400 mg Cap QD (Ph Ib) (N=6) | 800 mg Cap QD (Ph Ib) (N=7) | 200 mg Cap BID (Ph Ib) (N=4) | 400 mg Cap BID (Ph Ib) (N=12) | 600 mg Cap BID (Ph Ib) (N=5) | 200 mg Tab BID (Ph Ib) (N=7) | 400 mg Tab BID (Ph Ib) (N=8) | 400 mg Cap BID (Ph II) (N=53) | 400 mg Tab BID (Ph II) (N=47)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac disorder (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erysipelas (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Klebsiella infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Peritonitis bacterial (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 2
Pneumonia mycoplasmal (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Septic shock (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Tracheobronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood pressure decreased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peritumoural oedema (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intracranial pressure increased (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Spinal cord compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1 | 1
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 100 mg Cap QD (Ph Ib) (N=5) | 200 mg Cap QD (Ph Ib) (N=7) | 400 mg Cap QD (Ph Ib) (N=6) | 800 mg Cap QD (Ph Ib) (N=7) | 200 mg Cap BID (Ph Ib) (N=4) | 400 mg Cap BID (Ph Ib) (N=12) | 600 mg Cap BID (Ph Ib) (N=5) | 200 mg Tab BID (Ph Ib) (N=7) | 400 mg Tab BID (Ph Ib) (N=8) | 400 mg Cap BID (Ph II) (N=53) | 400 mg Tab BID (Ph II) (N=47)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 18 | 4
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 5 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 4 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Eye irritation (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0
Photopsia (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Visual acuity reduced (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 1 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 4
Constipation (Gastrointestinal disorders) | 3 | 2 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 5 | 11
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 3 | 4 | 1 | 1 | 3 | 7 | 15
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Duodenal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 3 | 1
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 3 | 6 | 2 | 1 | 1 | 5 | 3 | 7 | 26
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 3
Vomiting (Gastrointestinal disorders) | 2 | 3 | 2 | 7 | 1 | 1 | 1 | 2 | 3 | 10 | 10
Asthenia (General disorders) | 0 | 1 | 1 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 4
Chest discomfort (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Face oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 10 | 17
Generalised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 2 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 8 | 4
Oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 3
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1 | 1 | 4 | 2 | 3 | 2 | 15 | 21
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Peripheral swelling (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 3
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 1 | 1 | 2 | 4
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Eye infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Infected dermal cyst (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Localised infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 5 | 1
Paronychia (Infections and infestations) | 2 | 1 | 2 | 0 | 2 | 4 | 0 | 2 | 3 | 7 | 10
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 4
Hand fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 0 | 13 | 5
Amylase increased (Investigations) | 2 | 1 | 0 | 0 | 1 | 4 | 0 | 2 | 1 | 7 | 11
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 10 | 7
Bilirubin conjugated increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 0
Blood albumin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 2 | 4
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 5 | 0 | 0 | 0 | 8 | 4
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 3 | 1 | 2 | 0 | 9 | 8
Blood glucose increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood iron decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Blood phosphorus increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Crystal urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 5
Haemoglobin decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3 | 0
Lipase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 5 | 10
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Protein total increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Protein urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0
Urinary sediment present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine analysis abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Urine ketone body present (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 0
Urobilinogen urine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 2 | 0 | 4
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
White blood cells urine positive (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 2 | 1 | 4 | 1 | 1 | 3 | 3 | 3 | 13 | 19
Hyperamylasaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2 | 3 | 7 | 1 | 0 | 0 | 23 | 12
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 8 | 3
Hypochloraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 7 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 6 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1
Hypoproteinaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 5 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 4 | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Ligament pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 1 | 3
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 3 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 0 | 0 | 2 | 6 | 3
Dyskinesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Facial spasm (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 1 | 3 | 3 | 8
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 1
Nervous system disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Taste disorder (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 3 | 1 | 7 | 2
Azotaemia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Dysuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 5 | 2
Haemoglobinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1 | 1 | 3 | 3 | 0 | 1 | 14 | 8
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 2 | 1 | 4 | 1 | 1 | 2 | 3 | 9
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 8 | 2
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 4 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 1 | 0 | 1 | 0 | 4 | 1 | 0 | 5
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 2 | 5
Rash (Skin and subcutaneous tissue disorders) | 2 | 3 | 0 | 2 | 2 | 4 | 1 | 2 | 3 | 7 | 15
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.